CLINICAL TRIAL: NCT05508568
Title: A Performance Evaluation Study of Arquer's MCM5 Elisa Test (ADXBLADDER) to Aid in the Monitoring of Recurrence in Non-Muscle Invasive Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Arquer Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Arquer-US1
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Non-muscle invasive bladder cancer; MCM5; Biomarker; Urinary biomarker; Follow-up; Surveillance
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine sediment lysate samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Non-muscle invasive bladder cancer patients in follow-up: Patients with a previous diagnosis of non-muscle invasive bladder cancer, attending a urology clinic for the purposes of bladder cancer recurrence monitoring.
  Interventions: Diagnostic Test: ADXBLADDER

INTERVENTIONS:
Diagnostic Test: ADXBLADDER — ADXBLADDER is a non-invasive, qualitative ELISA utilising a combination of two monoclonal antibodies for the detection of MCM5 in urine sediment. It is intended to aid in the monitoring of bladder cancer recurrence in non-muscle-invasive bladder cancer patients. Participants will be asked to provide a full void urine specimen, which will be centrifuged before the urine sediment is lysed. The lysed sample will then be tested with ADXBLADDER.

SUMMARY:
The objective of this prospective, multi-centre study is to evaluate the performance of ADXBLADDER, a urine MCM5 ELISA test, as an aid in the detection of bladder cancer recurrence. Patients undergoing cystoscopic surveillance in non-muscle invasive bladder cancer (NMIBC) follow-up will be recruited and asked to provide a urine sample to be tested with ADXBLADDER. To assess the diagnostic accuracy of the test, the MCM5 results will be compared with the gold standard cystoscopy and pathology of resected tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with NMIBC in the previous 2 years, and are attending the urology clinic for standard of care/routine monitoring cystoscopy
* Patients 22 years of age or older
* Patients who, in the opinion of the Investigator, are suitable for standard urological investigations as part of normal clinical practice
* Patients who are, in the opinion of the Investigator, able to understand the purpose of the study and provide a full void urine specimen
* Patients who are able to give voluntary, written informed consent to participate in this study

Exclusion Criteria:

* Patients with known active (symptomatic) calculi within the urino-genitary system
* Patients who provide less than 10mL of full void urine
* Patients undergoing active treatment for interstitial cystitis
* Patients currently undergoing systemic chemotherapy or systemic immunotherapy or radiotherapy. Intravesical chemotherapy or immunotherapy (BCG) is allowed
* Patients who have previously been diagnosed with renal cancer, prostate cancer, Muscle Invasive Bladder cancer, an upper tract tumour, or CiS in the prostatic urethra
* Patients who have had urological instrumentation to the urinary tract within 14 days prior to the test
* Male patients undergoing active treatment for prostatitis

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cystoscopic surveillance for non-muscle invasive bladder cancer (NMIBC) follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity and negative predictive value (NPV) of ADXBLADDDER will be calculated to establish the diagnostic accuracy for the detection of bladder cancer recurrence. | Urine samples will be collected from participants immediately prior to cystoscopy and analysed for MCM5 within 6 months. Overall performance characteristics of ADXBLADDER will be established following study completion.
  The ADXBLADDER MCM5 results will be compared with the definitive diagnosis obtained by gold standard cystoscopy and pathological assessment of suspicious lesion(s) (where clinically indicated).

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ashish Kamat, Principal Investigator — M.D. Anderson Cancer Center
Locations (13):
- United States (13):
  - The Urology Center of Colorado, Denver, Colorado
  - Advanced Urology Institute, Daytona Beach, Florida
  - First Urology, Jeffersonville, Indiana
  - Michigan Institute of Urology, Troy, Michigan
  - New Jersey Urology, Mount Laurel, New Jersey
  - Associated Medical Professionals of NY, Syracuse, New York
  - Clinical Research Solutions, Cleveland, Ohio
  - MidLantic Urology, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas
  - Virginia Urology Center, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Spokane Urology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roupret M, Gontero P, McCracken SRC, Dudderidge T, Stockley J, Kennedy A, Rodriguez O, Sieverink C, Vanie F, Allasia M, Witjes JA, Colombel M, Sylvester R, Longo F, Montanari E, Palou J. Diagnostic Accuracy of MCM5 for the Detection of Recurrence in Nonmuscle Invasive Bladder Cancer Followup: A Blinded, Prospective Cohort, Multicenter European Study. J Urol. 2020 Oct;204(4):685-690. doi: 10.1097/JU.0000000000001084. Epub 2020 Apr 21. PMID 32314931
- [Background] Gontero P, Montanari E, Roupret M, Longo F, Stockley J, Kennedy A, Rodriguez O, McCracken SRC, Dudderidge T, Sieverink C, Vanie F, Allasia M, Witjes JA, Sylvester R, Colombel M, Palou J. Comparison of the performances of the ADXBLADDER test and urinary cytology in the follow-up of non-muscle-invasive bladder cancer: a blinded prospective multicentric study. BJU Int. 2021 Feb;127(2):198-204. doi: 10.1111/bju.15194. Epub 2020 Aug 29. PMID 32745350